CLINICAL TRIAL: NCT05231109
Title: The Effect of Vestibular Rehabilitation on Balance and Quality of Life in Patients With Bilateral Vestibular Hypofunction
Brief Title: Effect of Vestibular Rehabilitation in Patients With Bilateral Vestibular Hypofunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.53654
Record Dates: First submitted 2022-01-13; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2019-01

CONDITIONS: Individuals With Vestibular Hypofunction; Individuals Between the Ages of 18-65
Keywords: Bilateral vestibular hypofunction; Quality of life; Balance; Vestibular rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vestibular rehabilitation group (Other): Vestibular rehabilitation was performed. The following exercises were done with the patients: vestibular adaptation exercises, oculo-motor exercises, standing by changing the support area, the support surface and the arm positions, heel-toe walking, walking with head rotation, backward walking, counting on a soft surface with eyes open and closed, and dynamic balance exercises were taught to the patients. The exercise program was arranged 3 times a day for 6 months, and each exercise was 10 repetitions. The patients were called for physiotherapist control once every 2 weeks.
  Interventions: Other: vestibular rehabilitation

INTERVENTIONS:
Other: vestibular rehabilitation — Vestibular rehabilitation consisted of a total of 12 sessions, rearranged every 15 days. These exercises were prepared gradually to increase the vestibulo-ocular reflex and vestibulospinal reflex. The following exercises were done with the patients: vestibular adaptation exercises, oculo-motor exercises, standing by changing the support area, the support surface and the arm positions, heel-toe walking, walking with head rotation, backward walking, counting on a soft surface with eyes open and closed, and dynamic balance exercises were taught to the patients. The therapist gave the patients a home exercise program. It was emphasized that the exercises should be applied as 10 repetitions. After the session, the exercises shown to the patients were explained in written form and given as home exercises. They were also asked to do home exercises 3 times a day, 10 repetitions, for 15 days. Patients were re-evaluated before the treatment, at the 3rd month and after the 6th month.

SUMMARY:
Bilateral vestibular function is a heterogeneous chronic condition characterized by bilaterally decreased or absent function of vestibular organs, vestibular nerves, or both.1 Patients present with various symptoms such as oscillopsia, imbalance, visual vertigo, cognitive deficits, autonomic symptoms, and impaired spatial orientation. The aim of this study is to investigate the effectiveness of vestibular rehabilitation on balance, dynamic visual acuity and quality of life in patients with bilateral vestibular hypofunction. Twenty patients diagnosed with bilateral vestibular hypofunction by videonystagmography were included in the study. Balance Tests, Visual Analogue Scale, Dynamic Visual Acuity, Dizziness Disability Inventory for quality of life, computer modified for Sensory Interaction in Balance Clinical Test (MCTSIB) tests and Limits of Stability test, which provides evaluation of body movements, which are an important part of balance, in all directions. Evaluations were made at 3 and 6 months before treatment. Physiotherapy sessions were given at two-week intervals. According to the development of the patients, they were asked to perform a home exercise program with 10 repetitions 3 times a day.

DETAILED DESCRIPTION:
After the initial evaluations, the patients included in the study were included in the rehabilitation program. The rehabilitation program consisted of two phases. The first phase included patient education. All patients were planned to receive a verbal training for 30 minutes by the physiotherapist, including the definition of unilateral vestibular hypofunction, its importance, risk factors, ways of prevention, and recommendations for preventing falls. The second phase consisted of the vestibular exercise program. In this phase, vestibular adaptation exercises, oculo-motor exercises, standing by changing the support area, the support surface and the arm positions, heel-toe walking, walking with head rotation, backward walking, counting on a soft surface with eyes open and closed, and dynamic balance exercises were taught to the patients. The exercise program was arranged 3 times a day for 6 months, and each exercise was 10 repetitions. The patients were called for physiotherapist control once every 2 weeks. Patients were re-evaluated before the treatment, at the 3rd month and after the 6th month.

ELIGIBILITY:
Inclusion Criteria:

1. To be diagnosed with bilateral vestibular hypofunction by Videonystagmography test
2. To be between the ages of 18-75
3. To have communication and cooperation skills
4. To have no problems originating from the central nervous system
5. To have previously had ear infections, not having undergone surgery

Exclusion Criteria:

1. Having cognitive dysfunction
2. Presence of temporal bone pathologies detected by magnetic resonance imaging
3. Presence of other inner ear disorders that may cause dizziness and imbalance as determined by audiogram, tympanogram, and acoustic reflexes
4. Previous lower extremity injuries
5. The presence of central findings in Videonystagmography results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Static Posture Evaluation at 6 Months (Limits of Stability and modified for Sensory Interaction in Balance Clinical Test ) | 6 months
  With the limits of stability program on the balance device called Otometrics ICS Balance Platform, the body's final reaching points, the speed of movement, and direct control were evaluated, in 8 directions. Within this device, the modified for Sensory Interaction in Balance Clinical Test test was evaluated by showing areas of oscillation. Modified-CTSIB is a clinical test that is generally used as a semi-quantitative test measurement, and is scored according to the person's ability to perform various standing static positions.Before removing the patient on the device, the center of gravity is determined by entering the height and weight, and the patient visually sees the center of gravity when he/she gets on the balance platform. Then all tests are done according to this center of gravity.
Change from Baseline Dizziness Handicap Inventory at 6 Months | 6 months
  Dizziness Handicap Inventory was used to evaluate the quality of life of patients. This scale consists of 25 items that determine the aggravating factors of patients' dizziness and balance disorder, as well as emotional and functional outcomes in vestibular system diseases.

SECONDARY OUTCOMES:
Results of Dynamic Visual Acuity, Subjective Visual | 6 months
  The test was performed using the Snellen visual acuity chart. During the test, the patient was first asked where he read on the eye board on the wall while the head was fixed, and it was recorded. Then, while the patient's head was turned to the right and left rapidly 2 times per second, the patient was asked to continue reading on the eye board, and the answers were recorded.
Results of Dizziness Severity Scale, Subjective Visual | 6 month
  A 10-cm visual analog scale was used for evaluation. Patients were asked to rate the severity of dizziness on a scale of 0-10. It was explained that a score of "0" meant no dizziness at all, while a score of "10" indicated the presence of unbearable dizziness, and the patient was asked to mark the appropriate part.
Results of Tandem, Semi-tandem, Romberg and One-Leg Stance Test, Subjective Visual | 6 months
  For balance tests, tandem, semitandem, romberg, standing on one leg on hard ground, and standing on one leg on soft ground were evaluated with eyes open and eyes closed, and the second was recorded as seconds with a stopwatch. The test was considered completed in patients who could stand for 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Kılıç, master, Principal Investigator — PhD student; Z. Candan Algun, professor, Study Director — head of physical medicine and rehabilitaton department
Locations (1):
- Bağcılar Safa Hastanesi, Bağcılar, Yıldıztepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No